CLINICAL TRIAL: NCT05561374
Title: A Phase 1b Open-Label Study Investigating the Tolerability, Safety, and Pharmacokinetic Properties of Oral OKN-007 in Patients with Recurrent High-Grade Glioma
Brief Title: Study of Safety and Pharmacokinetic Properties of Oral OKN-007 in Patients with Recurrent High-Grade Glioma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Oblato, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OKN-007-OL-RMG-101
Record Dates: First submitted 2022-09-22; First posted 2022-09-30 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: High-grade Glioma; Oligodendroglioma; Astrocytoma; Glioblastoma Multiforme
MeSH Terms: conditions — Glioma; Oligodendroglioma; Astrocytoma; Glioblastoma | interventions — OKN 007; BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Low-dose OKN-007, two times a day (BID) (Experimental): Dose Escalation Cohort 1
  Interventions: Drug: Low-dose OKN-007, BID
- Low-dose OKN-007, three times a day (TID) (Experimental): Dose Escalation Cohort 2
  Interventions: Drug: Low-dose OKN-007, TID
- Mid-dose OKN-007, three times a day (TID) (Experimental): Dose Escalation Cohort 3
  Interventions: Drug: Mid-dose OKN-007, TID
- High-dose OKN-007, three times a day (TID) (Experimental): Dose Escalation Cohort 4
  Interventions: Drug: High-dose OKN-007, TID

INTERVENTIONS:
Drug: Low-dose OKN-007, BID — Participants will be administered low doses of oral OKN-007 two times a day daily in 28-day cycles.
  Arms: Low-dose OKN-007, two times a day (BID)
Drug: Low-dose OKN-007, TID — Participants will be administered low doses of oral OKN-007 three times a day daily in 28-day cycles.
  Arms: Low-dose OKN-007, three times a day (TID)
Drug: Mid-dose OKN-007, TID — Participants will be administered mid doses of oral OKN-007 three times a day daily in 28-day cycles.
  Arms: Mid-dose OKN-007, three times a day (TID)
Drug: High-dose OKN-007, TID — Participants will be administered high doses of oral OKN-007 three times a day daily in 28-day cycles.
  Arms: High-dose OKN-007, three times a day (TID)

SUMMARY:
This is a phase 1 open-label, multicenter study to investigate tolerability, safety and PK properties of oral OKN-007 in patients with recurrent high-grade glioma.

DETAILED DESCRIPTION:
This phase 1 open-label study is based on the traditional 3+3 design following the initial single-participant cohort to determine the maximum tolerated dose (MTD). Eligible participants will be enrolled each of the cohorts with escalated dose levels and administered the study drug OKN-007 orally daily in 28-day cycles: Cohort 1, Cohort 2, Cohort 3, Cohort 4. Participants may receive study treatment up to 2 years or until tumor progression, unacceptable toxicity, death, or patient withdrawal. The safety and pharmacokinetic properties of oral OKN-007 will be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed recurrent gliomas that were originally diagnosed as high-grade glioma (World Health Organization [WHO] Grade 3 or 4; astrocytoma, oligodendroglioma, or glioblastoma) by histopathology or molecular studies.
2. Progressive or recurrent gliomas documented by magnetic resonance imaging (MRI) no earlier than 180 days after first surgery for gliomas and no earlier than 90 days after completion of radiotherapy (applies to patients with first progression/recurrence only).
3. Patients must have medical records available documenting known histology or molecular and genetic information resulting from prior analyses, or tumor tissue samples available from prior glioma surgery or open biopsy for correlative research.
4. For patients with unresected recurrent tumor, unequivocal radiographic evidence of tumor progression by MRI as per the RANO criteria within 28 days prior to the first dose. These patients must have at least one measurable lesion per RANO.
5. No more than two prior lines of therapy for high-grade glioma (WHO Grade 3 or 4). The first-line therapy must include radiotherapy (minimum of 50 Gy; 34 Gy in elderly patients) with concomitant or adjuvant standard chemotherapy (temozolomide (TMZ), or procarbazine, lomustine and vincristine in patients with anaplastic oligodendroglioma).
6. Eastern Cooperative Oncology Group (ECOG) performance status <2.
7. Full recovery (grade ≤1) from the toxic effects of any earlier intervention and a minimum of 28 days from the last administration of any investigational agent that has not received regulatory approval for any indication at the time of registration.
8. Adequate renal, liver and bone marrow function without packed red blood cell/platelet transfusions within 4 weeks of the date of lab test during screening:

   * Leukocytes ≥3.0 × 10^9/L
   * Absolute neutrophil count (ANC) ≥1.5 × 10^9/L
   * Platelets ≥100 × 10^9/L
   * Hemoglobin ≥ 9.0 g/dL
   * Total bilirubin ≤1.5 × upper limit of normal (ULN), unless documented Gilbert's syndrome.
   * Aspartate transaminase/alanine transaminase ≤2.5 × ULN
   * Creatinine clearance ≥60 mL/min calculated as per Cockcroft-Gault equation.
9. Patients must be ≥18 years of age.
10. Life expectancy (as assessed by the Investigator) at least three months.
11. Patients must not have significantly diseased or obstructed gastrointestinal tract, malabsorption, uncontrolled vomiting or diarrhea, or inability to swallow oral medications.
12. Have provided written informed consent.
13. Patients must be willing to have multiple blood draws for PK analysis.
14. Female patients, of childbearing potential, must have a negative serum pregnancy test within 7 days prior to study treatment initiation and agree to use adequate contraception or practice sexual abstinence as the preferred and usual lifestyle of the patient during the study and for up to 120 days (4 months) after the last dose of study treatment.
15. Male patients with female partners of childbearing potential must, even if surgically sterilized, agree to practice effective barrier contraception and practice true abstinence.
16. Human immunodeficiency virus infected patients on effective antiretroviral therapy with undetectable viral load within 6 months prior to study registration are eligible for this trial.

Exclusion Criteria:

1. Prior malignancy (other than glioma) expected to require treatment within a 6-month period (except adequately treated basal cell carcinoma of the skin). Patients who had another malignancy in the past but have been free of active disease for more than 2 years, are eligible.
2. Have received treatment within the last 28 days with a drug that has not received regulatory approval for any indication at the time of study registration.
3. Have received chemotherapeutic agents (including TMZ) within 28 days or within 5 half-lives for non-cytotoxic agents (whichever is shorter) of study registration.
4. Serious concomitant systemic disorders, for example, abnormal electrocardiogram (ECG) indicative of cardiac disease (patients with Fridericia-corrected QT interval [QTcF] >480 msec.
5. Patients with abnormal sodium, potassium, or creatinine levels grade ≥2.
6. Inability to comply with protocol or study procedures.
7. Women who are pregnant or breastfeeding.
8. Patients who have received bevacizumab for recurrent glioblastoma or are planning to initiate treatment with bevacizumab for tumor necrosis.
9. Patients completing radiotherapy treatment less than 2 weeks prior to planned study treatment initiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability: Adverse events | From Day 1 to 30 days after the last treatment
  Safety and tolerability will be evaluated from adverse events as reported according to CTCAE version 5.0.
Pharmacokinetic profile: Maximum plasma concentration (Cmax) | Pre-dose, 2 hours, 4 hours, 5 hours, 6 hours, and 8 hours post-dose on Days 1 in Cycle 1 and 2; 5 hours post-dose on Day 5; Pre-dose, 5 hours post-dose on Day 8 in Cycle 1; Pre-dose on Days 1 of Cycle 3 and 4 (each cycle is 28 days)
  Maximum plasma concentration (Cmax) will be calculated using the actual sample collection times.
Pharmacokinetic profile: Time to Cmax (Tmax) | Pre-dose, 2 hours, 4 hours, 5 hours, 6 hours, and 8 hours post-dose on Days 1 in Cycle 1 and 2; 5 hours post-dose on Day 5; Pre-dose, 5 hours post-dose on Day 8 in Cycle 1; Pre-dose on Days 1 of Cycle 3 and 4 (each cycle is 28 days)
  Time to Cmax (Tmax) will be calculated using the actual sample collection times.
Pharmacokinetic profile: Area under the curve (AUC) | Pre-dose, 2 hours, 4 hours, 5 hours, 6 hours, and 8 hours post-dose on Days 1 in Cycle 1 and 2; 5 hours post-dose on Day 5; Pre-dose, 5 hours post-dose on Day 8 in Cycle 1; Pre-dose on Days 1 of Cycle 3 and 4 (each cycle is 28 days)
  Area under the curve (AUC) will be calculated using the actual sample collection times.
Pharmacokinetic profile: Half-life time (t1/2) | Pre-dose, 2 hours, 4 hours, 5 hours, 6 hours, and 8 hours post-dose on Days 1 in Cycle 1 and 2; 5 hours post-dose on Day 5; Pre-dose, 5 hours post-dose on Day 8 in Cycle 1; Pre-dose on Days 1 of Cycle 3 and 4 (each cycle is 28 days)
  Half-life time (t1/2) will be calculated using the actual sample collection times.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Providence Saint John's Cancer Institute, Santa Monica, California
  - Norton Healthcare, Louisville, Kentucky
  - Atrium Health Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina
  - The University of Oklahoma Health Sciences Center, Stephenson Cancer Center, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: No